CLINICAL TRIAL: NCT04325880
Title: Efficacy of Mirabegron Versus Tamsulosin Versus Solifenacin for Treatment of Ureteral Stents-Related Symptoms: a Randomized Controlled Trial
Brief Title: Efficacy of Mirabegron Versus Tamsulosin Versus Solifenacin for Treatment of Ureteral Stents-Related Symptoms
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AE 24320
Record Dates: First submitted 2020-03-24; First posted 2020-03-30 (Actual); Last update posted 2021-11-23 (Actual); Status verified 2021-11

CONDITIONS: Ureteral Stent; Stent Related Symptoms
Keywords: Ureteral stone; Ureteral stent; Stent related symptoms; Quality of life
MeSH Terms: conditions — Ureterolithiasis | interventions — mirabegron; Tamsulosin; Solifenacin Succinate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo arm (Placebo Comparator): Patients in this arm will receive a placebo formula
  Interventions: Drug: Placebo oral tablet
- Mirabegron arm (Active Comparator): Patients in this arm will receive Mirabegrone 50 mg once daily
  Interventions: Drug: Mirabegron 50 MG
- Tamsulosin arm (Active Comparator): Patients in this arm will receive tamsulosin o.4 mg once daily
  Interventions: Drug: Tamsulosin
- Solifenacin arm (Active Comparator): Patients in this arm will receive solifenacin 10 mg once daily
  Interventions: Drug: Solifenacin Succinate 10 MG

INTERVENTIONS:
Drug: Mirabegron 50 MG — Patients in this arm will receive Mirabegrone 50 MG once daily
  Arms: Mirabegron arm
Drug: Tamsulosin — Patients in this arm will receive Tamsulosin o.4 MG once daily
  Arms: Tamsulosin arm
Drug: Solifenacin Succinate 10 MG — Patients in this arm will receive Solifenacin Succinate 10 MG once daily
  Arms: Solifenacin arm
Drug: Placebo oral tablet — Patients in this arm will receive placebo oral tablet once daily
  Arms: Placebo arm

SUMMARY:
The primary objective of this prospective, single-centre randomized controlled trial is to assess the efficacy of three different drugs in treatment of ureteral stents related symptoms (Beta 3 adrenergic receptor agonist; Mirabegron 50mg) vs. (Alpha 1 adrenergic receptor antagonist; Tamsulosin 0.4mg) vs. (Anticholinergic; Solifenacin 10 mg) using validated symptoms questionnaires.

In addition, adverse events of the utilized medications will be monitored during study period as a secondary objective.

DETAILED DESCRIPTION:
Indwelling ureteral stents are specialized catheters designed to alleviate obstruction by maintaining the patency of the ureteral lumen and to splint the ureter by acting as a scaffold to promote organized tissue healing. (1)

Common issues associated with contemporary ureteral stents include stent-related pain, hematuria, dysuria, urgency, infection, and encrustation (2). Majority of patients (80%) reported one or more urinary symptoms with over 80% of patients experience stent-related pain that affects daily activities, 58% report reduced work capacity, and 32%report sexual dysfunction (2). In addition, as many as 32% of patients had ureteral stents removed sooner than anticipated because of these complications (3).

Considering this high prevalence of ureteral stent related symptoms (uSRS) among patients and its potential impact on quality of life (QoL), adequate management of these bothering symptoms was the point of research over the last decades (4).

The exact mechanism involved in uSRS is not yet known; however, many authors report that such symptoms are associated with ureteral spasms, urinary reflux attributable to ureteral stent, or trigonal irritation (5).

Different novel types of stents have been developed and evaluated to reduce uSRS; however, there is still controversy regarding their clinical application (6). Conversely, pharmacological therapy, including anticholinergics and alpha-blockers, remains the most effective option to manage uSRS (7).

The role of a-blockers in reducing uSRS involves reduction of bladder outlet resistance to alleviate flank pain in male patients with preexisting bladder outlet obstruction (BOO). It has been proposed that relaxing the distal ureter and irritation of the trigone decreases bladder outlet resistance and voiding pressure, thereby potentially decreasing the incidence of renal reflux and subsequent flank pain (8) . Otherwise, anticholinergic agents may have an effect on involuntary contractions of the bladder induced by the distal end of ureteral stents with subsequent relief of uSRS (9).

The above-mentioned drugs, however, are not easy to apply to some patients with co-morbidities because of the potential side effects. The most common medication-related complications of a-blockers are dizziness and orthostatic hypotension. Depending on the type of medication, medication-related adverse events are reported at a rate of 5% to 20% (10). In addition, anticholinergic agents have various adverse effects that decrease treatment compliance, such as dry mouth, constipation, blurred vision and dyspepsia (11).

Beta-3 agonist mirabegron is believed to be responsible for the relaxation of the detrusor smooth muscle during the storage phase (12). It helps relax the detrusor smooth muscle, and results in increased bladder capacity without any changes in micturition pressure, post-void residual urine volume, or voiding contractions.

Considering the function of mirabegron as a therapeutic agent for overactive bladder (OAB), mirabegron is assumed to be effective for relieving voiding symptoms attributable to uSRS (13).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 19-80 years)
* Undergo unilateral uncomplicated retrograde rigid ureteroscopy (URS) or retrograde intrarenal surgery (RIRS) with planned ureteral stent insertion.

Exclusion Criteria:

* Patients with neurogenic bladder, OAB syndrome, and neurological and psychiatric diseases
* Residual ureteral or renal stones after the procedure
* Preoperative febrile UTI
* pregnancy or breastfeeding
* Bilateral ureteroscopic surgery
* Single kidney
* Chronic kidney disease
* Cardiovascular or cerebrovascular disease
* Hepatic dysfunction
* History of pelvic surgery or irradiation
* History of bladder or prostate surgery
* Other acute medical conditions as acute gastroenteritis, osetoarthritis that might influence the patient QoL
* Preoperative indwelling of ureteral stent for relief of stone-related pain or sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in stent related symptoms using ureteral stent symptoms questionnaire (USSQ) | 4 weeks
  The effect of the assigned treatment on improvement of stent related symptoms will be assessed at the time of stent removal using ureteral stent symptoms questionnaire (USSQ)

SECONDARY OUTCOMES:
Adverse event of medications | 4 weeks
  Side effects of the assigned treatment will be monitored

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided